CLINICAL TRIAL: NCT04578470
Title: A Double Blinded Randomized Control Trial (RCT) to Evaluate the Effectiveness of Vitamin D Treatment in Lowering the Recurrence Rate of Benign Paroxysmal Positional Vertigo (BPPV) in Older Patients
Brief Title: Benign Paroxysmal Positional Vertigo (BPPV) in Older Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BPPV
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patient will also undertake a vitamin D and corrected calcium test. Based on the blood test results, the randomisation process and administration of Vitamin D treatment or placebo will be administered by unblinded team while the clinicians and the patients will remain blinded and will not be informed of their allocation within the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (No Intervention): Patients with replete VitaminD levels (≥30ng/ml) will be serving as a control in group C. Group C will not receive any Vitamin D intervention for the entire 12- month study period but will receive dietary interventions.
- Group A (Experimental): Group A will be prescribed Vitamin D supplementation in the form of daily 2000 IU cholecalciferol (two tablets)for 13 weeks, and daily1000 IU cholecalciferol(1tablet) for another 13 weeks and then treatment will be discontinued but dietary interventions will continue across the 12-month study period.
  Interventions: Drug: Vitamin D
- Group B (Placebo Comparator): Group B will be prescribed placebo of Vitamin D with two tablets daily for 13 weeks then 1 tablet daily for13 weeks then no treatment for 26 weeks but dietary interventions will continue across the 12-month study period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Daily 2000 IU cholecalciferol(two tablets) for 13 weeks,and daily 1000 IUcholecalciferol(1 tablet) foranother 13 weeks.
  Arms: Group A
Drug: Placebo — two tablets daily for 13weeks then 1 tablet daily for13 weeks
  Arms: Group B

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is the most common cause of vertigo in older adults (Parham & Kuchel, 2016). It is caused by dislodged otoconia, which fall from the utricular macula into the semicircular canals causing them to move through the canals with the effect of gravity (Parnes et al., 2003). Treatment of BPPV is primarily with Canalith Repositioning Procedure (CRP) with more than 80% success rates. However, BPPV can recur in 10-20% of the time and in some long-term follow-up studies reporting up to 50% recurrence rates (Fife et al., 2008). Despite BPPV being considered a benign self-limiting condition, it has far reaching physical and psychosocial consequences for the geriatric population such as injuries from falls precipitated by vertiginous attacks and fear of unexpected vertigo leading to restriction of daily activities and functional decline (Balatsouras et al., 2018; Kao et al., 2009). Studies have shown that the 1-year prevalence of individuals with BPPV attacks rises steeply with age, with the cumulative (lifetime) incidence of BPPV reaching almost 10% by the age of 80 (Parham & Kuchel, 2016). Aging has also been shown to be a primary risk factor for idiopathic BPPV, with events such as prolonged bed rest postulated for being a trigger for BPPV (Parham & Kuchel, 2016). BPPV is also noted to be underreported in the elderly mainly due to the different manifestations such as less rotatory vertigo and more nonspecific dizziness and instability, with consecutive examinations in geriatric population revealing that 9% of elderly have unrecognized BPPV (Oghalai et al., 2000). Given the increased prevalence and severe implications of BPPV on there is a strong impetus for this study to lower the recurrence of BPPV in this vulnerable older population.

DETAILED DESCRIPTION:
The study aims to investigate whether Vitamin D supplementation with diet, or diet alone combined with CRP (standard clinical care) can reduce recurrence of BPPV and if there is any improvement in the patient's functional ability, postural stability and prevalence of falls.

* Group A will be prescribed Vitamin D supplementation in the form of daily 2000 IU cholecalciferol (two tablets) for 13 weeks, and daily 1000 IU cholecalciferol(1 tablet) for another 13 weeks and then treatment will be discontinued but dietary interventions will continue.
* Group B will be prescribed placebo of Vitamin D with two tablets daily for 13 weeks then 1 tablet daily for 13 weeks then no treatment for 26 weeks but dietary interventions will continue.
* Group C will not receive any Vitamin D intervention for the entire 12- month study period but will receive dietary interventions.

The same day, patients will be grouped according to their Vitamin D status. Patients who are Vitamin D deplete (<30ng/ml) will be randomised into groups A or B.

Randomisation will be undertaken by the unblinded team, who will allocate randomly generated treatment using sealed opaque envelopes. The unblinded team will open the sealed envelope and the patient will be allocated to a group. The patient will not be informed of the treatment regime. Patients with replete Vitamin D levels (≥30ng/ml) will be serving as a control in group C. All clinical investigators will be blinded to the group assignments.

Unblinding can be undertaken for urgent clinical need, for example, fall with hip fracture requiring surgical intervention and high dose replacement of Vitamin D prior to initiation of bisphosphonate or other osteoporosis treatment.

All request for unblinding will be made to the unblinded team investigator to determine the need for unblinding prior to release of unblinded information. However, the dosing chosen for the study would permit the patient to have treatment with clinically needed high doses of vitamin D and continue on the study treatment without risk of hypervitaminosis D. The anonymous google survey undertaken indicated that some clinicians will use high dose replacement at the same time as maintenance dosing. Any cases that require unblinding will be discussed with the unblinded Investigator before the unblinding takes place but the outcome of the unblinding will not be communicated to the clinical team to allow the study assessments to continue.

All Groups (A, B, C) will receive dietary interventions across the 12- month study period and will be scheduled dietitian clinics to attend. Before their clinics, all patients will be issued instructions by the dietitian to record their dietary habits via a 3-day food record (3DFR- Appendix 4) and to send their 3DFR to the dietitian through mail or email, at least 5 days prior to their scheduled dietitian review. Patients will be provided a unique patient identification number in the study and will be asked to use this number in place of personal particulars when sending in their 3DFR. In the event that patients are unable to send in their 3DFR before their appointment, they will be asked to bring it on the day of the review itself.

1-2 weeks appointment All Groups (A, B, C) will be scheduled an ENT review in 1-2 weeks as routine clinical care for patients following CRP. Alongside this ENT review, they will also receive a referral to the dietitian clinic at this routine clinical visit for assessment of their dietary habits. ENT clinic will test all patients for efficacy of CRP treatment. Dietitian's clinic will provide assessment of patients' dietary habits from their 3DFR, provide counselling on dietary habits as well as take anthropometric measurements such as height, weight and BMI.

3rd month tele- consult All Groups (A, B, C) will receive a call from the audiologist who will check on BPPV recurrence with specific questions from the Shortened Dizziness Handicap Inventory Questionnaire (SDHIQ).

6th month appointment All Groups (A, B, C) will return for an audiologist review and dietitian review. At the audiologist review, patients will answer questions relating to BPPV recurrence, undergo Dix Hallpike test to check for recurrence of BPPV and balance and functional assessment in the form of Gans SOP, SPPB, BI and CFS. Patients from Group A and B will also be required to bring in their prescribed medications for a final pill count in order to check for compliance (performed by unblinded team). At the dietitian review, there will be assessment of the patient's dietary habits from their 3DFR (which is to be submitted 5 days prior to visit), counselling on dietary habits and taking of anthropometric measurements such as height, weight and BMI.

9th month tele- consult All Groups (A, B, C) will receive a call from the audiologist who will check on BPPV recurrence with specific questions from the SDHIQ.

12th month appointment All Groups (A, B, C) will return for the final audiologist review and dietician review. At the audiologist review, all patients will answer questions relating to BPPV recurrence and undertake a Dix Hallpike test to check for recurrence of BPPV. The audiologist will also administer balance and functional assessment in the form of Gans SOP, SPPB, BI and CFS for comparison with start of study. All groups will undertake a final serum vitamin D3 test and corrected calcium measurements. At the dietitian review, there will be assessment of the patient's dietary habits from their 3DFR (which is to be submitted 5 days prior to visit), counselling on dietary habits and taking of anthropometric measurements such as height, weight and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >/=50 with a history suggestive of idiopathic BPPV, supported by a positive Dix Hallpike test. The study is to be undertaken in older patients hence the age criteria.
* Cognisant or mild neurocognitive impairment (AMT ≥7) to ensure the patient can provide informed consent.
* Both male and female participants will be recruited.

Exclusion Criteria:

* Patients with identified neurological causes of giddiness
* Patients with major neurocognitive impairment (severe dementia)
* Patients with sarcoidosis, metastatic disease (lymphoma, multiple myeloma), parathyroid disorders.
* Patients with diagnosed osteoporosis or osteopenia who are currently on high dose treatment (50,000 IU/week)
* Patients with significant cervical-spinal radiculopathy, spondylolisthesis, lordosis or kyphosis that will affect ability to carry out CRP
* Patients with disorders causing fat malabsorption (Short gut syndrome, Celiac disease) that will affect dietary absorption of Vitamin D
* Patients with Myasthenia Gravis
* Patients with unexplained hypercalcaemia
* Pregnant women (although this is extremely unlikely in age >/=50)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduce the recurrence rate of BPPV | 2 Years
  To determine if Vitamin D replacement in those deplete with Vitamin D, combined with dietary interventions, will reduce exacerbations of BPPV and thereby result in functional improvement.
Delay time to onset of recurrent episodes of BPPV | 2 Years
  To determine if Vitamin D replacement in those deplete with Vitamin D, combined with dietary interventions, will reduce exacerbations of BPPV and thereby result in functional improvement.